CLINICAL TRIAL: NCT05565820
Title: Treatment of Infestation With Pediculus Humanus Capitis in the Community Using a leave-in Spray: A Prospective, Randomised Controlled Study
Brief Title: A Study to Evaluate the Efficacy and Safety of a Leave-in Spray in Subjects With Head Lice Infestation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alliance Pharmaceuticals (Industry)
Collaborators: South Florida Family Health and Research Centers (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALLI010-0021
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Pediculosis Capitis; Lice Infestations; Head Lice
Keywords: Phthiraptera; Pediculus humanus Capitis; Pediculidae; Parasitic Diseases; Human Head Louse; Pediculi; Nits; Homeopathy; Homeopathic Pharmacopoeias; Homeopathic Formularies; Insecticides; Parasitology
MeSH Terms: conditions — Lice Infestations; Parasitic Diseases

STUDY DESIGN:
Intervention Model Description: Parallel group design with participants randomised, Randomly assign subjects to treatment or control group based on infestation severity alternation system, to Vamousse Spray 'n' Go or 1% Permethrin control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vamousse Spray 'n' Go (Experimental): Clinical staff will apply Vamousse Spray 'n' Go during the baseline visit (Day 0) to fully coat the hair and scalp. The treatment will be left on for 8 hours, then standard at home shampoo will be used and rinsed off with warm water, followed by combing. At day 7, if live lice are still present, a repeat treatment will be administered.
  Interventions: Other: Vamousse Spray 'n' Go
- Nix Creme Rinse Lice Treatment (Active Comparator): During the baseline visit (Day 0) clinical staff will first shampoo the hair and scalp using regular shampoo. They will then thoroughly rinse and towel dry the hair and scalp, and allow hair to air dry for a few minutes. Staff will shake Nix Creme Rinse Lice Treatment (1% permethrin lotion) well before applying, they will then proceed to thoroughly wet the hair and scalp with the lotion, being sure to cover the areas behind the ears and on the back of the neck. After allowing the lotion to remain in place for 10 minutes, they will rinse the hair and scalp thoroughly and dry with a clean towel. At day 7, if live lice are still present, a repeat treatment will be administered.
  Interventions: Drug: Nix Creme Rinse Lice Treatment

INTERVENTIONS:
Other: Vamousse Spray 'n' Go — Pediculicide for topical application, active ingredient Natrum Muriaticum 2X (HPUS).
  Arms: Vamousse Spray 'n' Go
Drug: Nix Creme Rinse Lice Treatment — 1% permethrin lotion for topical application.
  Arms: Nix Creme Rinse Lice Treatment

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Vamousse Spray 'n' Go, compared to a 1% Permethrin control shampoo, in the treatment of head lice.

DETAILED DESCRIPTION:
This is a Study to Evaluate the Safety and Efficacy of Alliance Pharmaceutical Product in Subjects Infested with Pediculosis Capitis. The subject population includes healthy male and female subjects aged 2 years and up who are infested with Pediculus humanus capitis. Household members infestation with an active head lice, defined as at least 1 live louse (adult and/or nymph) present on the scalp and/or hair as determined by a trained evaluator, will receive treatment with study product at baseline.

The planned overall sample size for this clinical trial is approximately n=58 subjects, equally divided between treatment and control groups. Potential subjects will be screened for eligibility and if eligible to participate, their infestation level will be rated. Eligible subjects at each infestation level will be assigned alternately to the treatment or control group to ensure that the two groups have approximately equal representations of infestation severity levels. Level of infestation will be rated as heavy, moderate or light described by how quickly lice were found during combing: heavy infestation = >1 louse with one stroke of the comb; moderate infestation =1 louse with one stroke of the comb; light infestation = first louse found only after several strokes of the comb.

Randomly assign subjects to treatment or control group based on infestation severity alternation system (i.e., randomly assign pairs of equal severity levels to treatment and control groups, a form of stratified random sampling) to achieve balanced representation of severity in the two groups.

After assignment to a study group, each eligible subject will receive the application of either the Alliance Pharmaceutical Product Vamousse Spray 'n' Go drug or the Permethrin-based control drug. Infested household members will be treated with the Vamousse Spray 'n' Go or Permethrin lotion on-site (i.e., the household members should be assigned to the same treatment as the index case). During the baseline visit (Day 0), the Investigator and clinical staff members will record subject's demographics; elicit informed consent; obtain medical history; review concomitant medication to identify any prohibited therapies the subject may be receiving; collect vital signs; conduct visual assessment of head lice, specifically counting live lice and nits with stages noted, using a 15 inch led 5x magnifying procedure lamp and if needed for confirmation, laboratory microscopes; perform physical examination; assess local skin/ scalp irritation; assess ocular irritation; perform urine pregnancy test on females; and conduct an adverse event assessment.

At day 7, if live lice are still present, a repeat treatment will be administered. After day 7 if a subject reports clear signs of infestation ( i.e., the presence of live lice), they will be regarded as a treatment failure and they will be offered treatment with an alternative product (viz., Vamousse Mousse ) by clinical staff.

For the treatment group, Clinical staff will apply Vamousse Spray 'n' Go to fully coat dry hair and scalp, avoiding the eyes and mucus membranes. The Treatment will be left on the hair and scalp for 8 hours, then standard at home shampoo and rinsed off with warm water, followed by combing. The Treatment spray bottle is intended for a single use although it contains a sufficient quantity for two treatments. All household members will be instructed on an overall lice management program, which includes:

* Wash (in hot water) or dry-clean all recently worn clothing, hats, used bedding and towels.
* Wash (in hot water) personal care items such as combs, brushes and hair clips.
* Record time and date product shampoo/rinse 8 hours post treatment

For the control group, Clinical staff will first shampoo the hair and scalp using regular shampoo. They will then thoroughly rinse and towel dry the hair and scalp, and allow hair to air dry for a few minutes. Shaking the permethrin lotion well before applying, they will proceed to thoroughly wet the hair and scalp with the permethrin lotion, being sure also to cover the areas behind the ears and on the back of the neck. After allowing the lotion to remain in place for 10 minutes, they will then rinse the hair and scalp thoroughly and dry with a clean towel.

The site will provide Subject with lice management instructions. Subjects will return for post-baseline visits assessments at Day 2, Day 7, and Day 14.

Day 2: The Investigator and medical staff will collect medical history, collect vital signs, perform physical examination, scalp irritation assessment, ocular irritation assessment and adverse events assessment, perform a visual assessment for the presence or absence of head lice, (Lice will be counted, each stage examined and noted live or dead; 15in led 5x magnifying procedure lamp or laboratory microscopes are used for confirmation if needed, Without clipping hair strands, nits will also be examined, each stage examined and noted hatched or unhatched), and adverse events assessment Urine pregnancy testing will be performed on each Visit, with interim visits confirming pregnancy has not occurred through questioning participating subject and legal guardian.

Day 7: The Investigator and medical staff will collect medical history, collect vital signs, perform a physical examination, assess scalp irritation, assess ocular irritation and adverse events, perform a visual assessment for the presence of head lice (lice will be counted, each stage identified, and noted live or dead; 15in led 5x magnifying procedure lamp or laboratory microscopes will be used for confirmation if needed; without clipping hair strands, nits will also be examined, each stage examined, and noted hatched or unhatched). Urine pregnancy testing of females will be performed on each visit, with interim visits confirming pregnancy has not occurred through questioning participating subject and legal guardian. If, at day 7, live lice are still present, a repeat Vamousse Spray 'n' Go or Permethrin (depending on study group) shampoo treatment will be administered.

Day 14: The Investigator and medical staff will collect medical history, concomitant and prohibited medication review, perform vital signs, urine pregnancy testing if applicable, perform physical examination, record local application site reactions, ocular irritation assessment, perform a visual assessment for the presence of head lice (lice will be removed, counted, each stage examined and noted live or dead; 15 inch led 5x magnifying procedure lamp or laboratory microscopes are used for confirmation; nits will also be removed by clipping hair strands, examined, each stage counted, and noted as hatched or unhatched) and adverse events assessment. By day 14 if a subject reports clear signs of infestation (i.e., the presence of live lice) they will be regarded as a treatment failure and will be offered treatment with an alternative product (Vamousse Mousse) by clinical staff.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have an active head lice infestation defined as: at least 1 live lice (adults and/or nymphs) present on the scalp and/or hair, as determined by a trained evaluator.
* Subjects must be at least two (2) years of age through 75 years of age, presenting with an active head lice infestation.
* Subject is male or female.
* Subject is in good general health based on medical history.
* Each subject must have an appropriately signed Informed Consent agreement. A caregiver must sign an Informed Consent agreement for children not old enough to do so. Children 6-17 years of age will be administered a child's Assent Form.
* The caregiver of a subject must be willing to allow all household members to be screened for head lice. If other household members are found to have an active head lice infestation, they must be willing and able to participate in receiving study product or Standard of Care.
* Subject agrees not to use any other form of lice treatments (commercial, community-anecdotal, or mechanical/manual) while participating in the study.
* Following application of the test product, subject agrees not to shampoo, wash or rinse their hair or scalp until 8-hour post-treatment time has been reached and documented.
* Subject agrees not to cut or chemically treat their hair while participating in the study.
* Subject agrees to follow all study instructions, including attending all follow-up appointments.
* Female subjects of childbearing potential must be willing to have a urine pregnancy test prior to inclusion in this study.

Exclusion Criteria:

* History of irritation or sensitivity to Nature Muriaticum 2X (HPUS) or Vamousse Spray 'n' Go or the components, pediculicides or hair care products.
* Presentation at the treatment site with visible skin/scalp condition(s) that are not attributable to head lice infestation, such as an erythema score and atopic dermatitis that is >2, blisters, vesicles which, in the opinion of the investigative personnel or medical monitor, will interfere with safety and/or efficacy evaluations.
* Presentation at the treatment site with eczema or atopic dermatitis.
* Treatment for head lice (Over the Counter, home remedy and/or Prescription) in the last 30 days.
* Any condition or illness that, in the opinion of the investigator, may compromise the objective of the protocol.
* Subject is receiving any other treatment which, in the opinion of the investigator or medical monitor, may interfere with the study results.
* Females (including caregivers who come in contact with the investigational product) who are pregnant, nursing or planning a pregnancy which could include household subjects. If a household has a pregnant female who has an active case of lice, the entire household is excluded from participation and provided Standard of Care.
* Household members of child-bearing potential, including subjects, and unwilling to use an adequate method of contraception for the duration of the study. Adequate methods of contraception include: abstinence, vasectomised partner, oral birth control pills, birth control injections or patches, intra uterine devices, condoms with a spermicidal jelly or a diaphragm with spermicidal jelly, surgical sterilisation. Subjects and/or caregivers will be considered non-child-bearing if the following has occurred: full hysterectomy or bilateral oophorectomy is considered surgically sterile. Tubal ligation is not considered equivalent to female sterilisation.
* Participation in a previous investigational drug study within the past 30 days.
* Does not understand the requirements for study participation and/or may likely exhibit poor compliance, in the opinion of the investigator.
* Does not have a known household affiliation with their household members (i.e., do not stay in one household consistently, sleeping at one place several nights and then at another place or location). Household is defined as living in a shared area or space (for example the same house of apartment unit).

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-03-12 (Actual); Study Completion 2023-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susel L Gonzalez Acosta, APRN, Principal Investigator — South Florida Family Health and Research Centers
Locations (1):
- South Florida Family Health and Research Centers, LLC., Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barker SC, Burgess I, Meinking TL, Mumcuoglu KY. International guidelines for clinical trials with pediculicides. Int J Dermatol. 2012 Jul;51(7):853-8. doi: 10.1111/j.1365-4632.2011.05446.x. PMID 22715834
- [Background] Birkemoe T, Lindstedt HH, Ottesen P, Soleng A, Naess O, Rukke BA. Head lice predictors and infestation dynamics among primary school children in Norway. Fam Pract. 2016 Feb;33(1):23-9. doi: 10.1093/fampra/cmv081. Epub 2015 Oct 28. PMID 26511728
- See also: Head Lice Infestation: Developing Drugs for Topical Treatment - Guidance for Industry. U.S. Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research October 2016 — https://www.fda.gov/regulatory-information/search-fda-guidance-documents/head-lice-infestation-developing-drugs-topical-treatment-guidance-industry

RESULTS

PARTICIPANT FLOW:
Groups:
- Vamousse Spray 'n' Go: 1. Recruitment Details:
     Upon arrival at the clinic, lice-infested patients and their household members were screened for eligibility against the inclusion and exclusion criteria. Those in each household who passed the screening were assigned to one of the two treatment groups through a reversing alternation assignment procedure.
  2. Type of Units Assigned:
     Vamousse Spray 'n' Go Treatment Group: members of this group were treated at baseline and, if live lice were found, again at Day 7 subsequent to baseline with the Vamousse Spray 'n' Go product, which is a pediculicide for topical application, having as its active ingredient Natrum Muriaticum 2X (HPUS).
  3. Periods:
     A. Baseline to Day 7 Assessment 1) Completed 41 of the 43 subjects in this group completed this period. 2) Not Completed 2 subjects in this group dropped out of the study prior to the Day 7 assessment. B. Baseline to Day 14 Assessment 1) Completed 41 of the original 43 subjects in this group completed this period. 2) Not Completed 2 subjects in this group dropped out of the study prior to the 14th day after baseline.
  4. Reasons Not Completed A. Reason Not Completed Type 1) Subject #16: Withdrawal by subject 2) Subject #17: Withdrawal by subject B. Reason Not Completed Data Withdrawal by subject: N = 2
- Nix Creme Rinse Lice Treatment: 1. Recruitment Details:
     Upon arrival at the clinic, lice-infested patients and their household members were screened for eligibility against the inclusion and exclusion criteria. Those in each household who passed the screening were assigned to one of the two treatment groups through a reversing alternation assignment procedure.
  2. Type of Units Assigned:
     Nix Creme Rinse Lice Treatment Group: members of this group were treated at baseline and, if live lice were found, again at Day 7 subsequent to baseline with the Nix Creme Rinse Lice Treatment product, which is a pediculicide topical application having as its active ingredient permethrin at 1% concentration.
  3. Periods:
     A. Baseline to Day 7 Assessment 1) Completed 15 of the 15 subjects in this group completed this period. 2) Not Completed No subjects in this group dropped out of the study prior to the Day 7 assessment. B. Baseline to Day 14 Assessment 1) Completed 15 of the original 15 subjects in this group completed this period. 2) Not Completed No subjects in this group dropped out of the study prior to the 14th day after baseline.
  4. Reasons Not Completed No subjects in this treatment group failed to complete the study.
Period: 2 Day Treatment Effectiveness
Arm/Group | Vamousse Spray 'n' Go | Nix Creme Rinse Lice Treatment
Started | 43 | 15
Completed | 43 | 15
Not Completed | 0 | 0
Period: 7 Day Treatment Effectiveness
Arm/Group | Vamousse Spray 'n' Go | Nix Creme Rinse Lice Treatment
Started | 43 | 15
Completed | 41 (The reason why the number of subjects in the Vamousse group who started the 7 day period is greater than the number of subjects who ended the 2 day period is that the periods are not consecutive but rather overlapping. Both periods started at Day 1 and had the same number of subjects at Day 1: 43 in the Vamousse Group (and 15 in the Permethrin group). Two subjects in the Vamousse Group withdrew from the study immediately after the Day 2 assessment and were not involved in the Day 7 assessment.) | 15
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: 14 Day Treatment Effectiveness
Arm/Group | Vamousse Spray 'n' Go | Nix Creme Rinse Lice Treatment
Started | 43 (The reason why the number of subjects in the Vamousse group who started the 14 day period is greater than the number of subjects who ended the 7 day period is that the periods are not consecutive but rather overlapping. Both periods started at Day 1 and had the same number of subjects at Day 1: 43 in the Vamousse Group (and 15 in the Permethrin group). Two subjects in the Vamousse Group withdrew from the study immediately after the Day 2 assessment and were not involved in the Day 14 assessment.) | 15
Completed | 41 | 15
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: The pattern of infestation levels of the primary participant in each household and the sizes of the households that were encountered in the sequential enrollment process resulted in an imbalance between the numbers of participants in the two treatment groups by the time that the study total of 58 participants was reached. Resources did not permit further enlargement of the sample to reduce this imbalance, but the power of the study to detect the difference that occurred remained high at .95.
Groups:
- Vamousse Spray 'n' Go: The Vamousse Spray 'n' Go group is defined as the group of lice infected subjects who were treated with the Vamousse Spray 'n' Go product at baseline and if needed, on Day 7 following baseline. Treatment with this product consisted of fully coating the hair and scalp with the product, leaving it on for 8 hours and then shampooing at home by the subject with the subject's usual shampoo, and rinsed off with warm water followed by combing.
- Nix Creme Rinse Lice Treatment: The Nix Creme Rinse Lice Treatment group is defined as the group of lice infected subjects who were treated with the Nix Creme Rinse Lice Treatment at baseline and if needed, on Day 7 following baseline. Treatment with this product consisted of the clinical staff first shampooing the subject's hair and scalp using regular shampoo and then thoroughly rinsing and towel drying the person's hair and scalp. After allowing the hair to air dry for a few minutes, they then thoroughly wet the subject's hair and scalp with the Nix Creme Rinse Lice Treatment lotion, being sure to cover the areas behind the ears and on the back of the neck.The lotion was allowed to remain in place for 10 minutes, after which the hair and scalp were thoroughly rinsed and dried with a clean towel.
- Total: Total of all reporting groups
Arm/Group | Vamousse Spray 'n' Go | Nix Creme Rinse Lice Treatment | Total
Number analyzed (Participants) | 43 | 15 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28 | 12 | 40
  Between 18 and 65 years | 15 | 3 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.72 (14.27) | 13.93 (13.87) | 17.48 (14.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 14 | 53
  Male | 4 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Hispanic | 43 | 15 | 58
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43 | 15 | 58
Count of live lice [Number; unit: live lice] — The count of live lice consisted of the number of live adult and nymph lice found anywhere above the shoulders on the subject.
  live lice | 1270 | 288 | 1558

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Are Completely Free of Live Lice
Description: The total numbers of subjects in each group free of live lice at Days 2, 7, and 14, where 'live lice free" is defined as no presence of live adult or nymph lice. Zero subjects in each group were free of live lice at baseline. Since the two groups differed substantially in size, the numbers of live lice free subjects in each group at Days 2, 7, and 14 were transformed for analytical purposes to proportions of the respective group's participant totals on the respective days in order to achieve a metric that reflects commensurate degrees of difference between the two groups.
Time Frame: 2, 7, and 14 days from baseline
Population: The 58 subjects who completed one or more of the three post-baseline assessments.
Measure: Number; unit: proportion of subjects free of live lice
Arm/Group | Vamousse Spray 'n' Go | Nix Creme Rinse Lice Treatment
Number analyzed (Participants) | 43 | 15
proportion of subjects free of live lice
  Baseline proportion | 0.00 | 0.00
  Day 2 proportion | .535 | .200
  Day 7 proportion: number analyzed (Participants) | 41 | 15
  Day 7 proportion | .415 | .067
  Day 14 proportion: number analyzed (Participants) | 41 | 15
  Day 14 proportion | .683 | .400
Statistical Analysis 1: Comparison: Vamousse Spray 'n' Go vs Nix Creme Rinse Lice Treatment; Null hypothesis: At Day 2 the proportion of lice free subjects in the Vamousse Spray 'n' Go group does not exceed that in the Nix Creme Rinse Lice Treatment group. The null hypothesis is one-tailed. However, for consistency with the practice of reporting conservative p-values in clinical studies, the two-tailed p-value will be reported; Test type: Superiority; p = .025, Z-test for difference in proportions — Alpha: .05; Z: 2.246 Cohen's d: .590; difference in proportions = -.335, Standard Error of Mean .149 — Direction of comparison: Vamousse Day 2 proportion of live lice - Nix Day 2 proportion of live lice
Statistical Analysis 2: Comparison: Vamousse Spray 'n' Go vs Nix Creme Rinse Lice Treatment; Null hypothesis: At Day 7 the proportion of lice free subjects in the Vamousse Spray 'n' Go group does not exceed that in the Nix Creme Rinse Lice Treatment group. The null hypothesis is one-tailed. However, for consistency with the practice of reporting conservative p-values in clinical studies, the two-tailed p-value will be reported; Test type: Superiority; p = .014, Z-test for difference in proportions — Alpha: .05; Z 2.469 Cohen's d .660; Difference in proportions = .348, Standard Error of Mean .141 — Direction of comparison: Vamousse Day 7 proportion live lice free - Nix Day 7 proportion live lice free
Statistical Analysis 3: Comparison: Vamousse Spray 'n' Go vs Nix Creme Rinse Lice Treatment; Null hypothesis: At Day 14 the proportion of lice-free subjects in the Vamousse Spray 'n' Go group does not exceed that in the Nix Creme Rinse Lice Treatment group. The null hypothesis is one-tailed. However, for consistency with the practice of reporting conservative p-values in clinical studies, the two-tailed p-value will be reported; Test type: Superiority; p = .054, Z-test for difference in proportions — Alpha: .05; Z: 1.920 Cohen's d: .513; Difference in proportions = .283, Standard Error of Mean .147 — Vamousse Day 14 proportion live lice free - Nix Day 14 proportion live lice free

2. Secondary Outcome: Proportion of Change in Total Number of Live Adult Lice and Nymphs From the Baseline
Description: The counts of live lice at Days 2, 7, and 14 for were subtracted from the respective each participant's baseline count for the respective day. The resulting raw differences were transformed for analytical purposes to proportions of the respective participant's baseline live lice count in order to achieve a metric that reflected commensurate degrees of change, the means of which could be compared between the two groups for each interval from baseline. All proportions of change from baseline are negatively signed to reflect a reduction in the count from baseline, which occurred for both groups on all 3 post-baseline assessment days.
Time Frame: 2, 7, and 14 days from baseline
Population: All subjects who had completed one or more of the three assessments during the 14 day post-baseline portion of the study.
Measure: Mean (Standard Deviation); unit: proportion of change in number live lice
Arm/Group | Vamousse Spray 'n' Go | Nix Creme Rinse Lice Treatment
Number analyzed (Participants) | 43 | 15
proportion of change in number live lice
  Day 2 proportion of change from baseline | -.859 (.225) | -.564 (.424)
  Day 7 proportion of change from baseline: number analyzed (Participants) | 41 | 15
  Day 7 proportion of change from baseline | -.762 (.666) | -.549 (.370)
  Day 14 proportion of change from baseline: number analyzed (Participants) | 41 | 15
  Day 14 proportion of change from baseline | -.926 (.177) | -.691 (.386)
Statistical Analysis 1: Comparison: Vamousse Spray 'n' Go vs Nix Creme Rinse Lice Treatment; Null hypothesis: At Day 2 the mean proportion of decrease from Day 0 in the number of live lice in the Vamousse group does not exceed that in the Nix group. The distribution of the Day 0 to Day 2 change proportions deviated significantly from normality by the Shapiro-Wilk test for both the Vamousse and combined samples. However, the t-test is robust to such departures from normality for samples of this size and was used to compare the two groups on the mean change proportions; Test type: Superiority — To check on the effect of the non-normality of the change proportions, the nonparametric Mann-Whitney test was also performed. The null hypothesis is one-tailed. However, for consistency with the practice of reporting conservative p-values in clinical studies, the two-tailed p-value will be reported; p = .020, t-test, 2 sided — Alpha = .05 t: 2.567 df (adjusted, see comment below): 16.83 Mann-Whitney Z: 2.830 p(2-tailed) of Mann-Whitney Z: .005 Cohen's d = 1.023; Degrees of freedom for the t-test were adjusted for inequality of variances between the groups using the Satterthwaite correction: df(adj) = 16.83; Mean Difference (Final Values) = .295, 95% CI 2-sided [.052 to .537], Standard Error of Mean .1148 — Direction of comparison: Vamousse prop. reduction in live lice count from Day O - Nix prop. reduction in live lice count from Day O
Statistical Analysis 2: Comparison: Vamousse Spray 'n' Go vs Nix Creme Rinse Lice Treatment; Null hypothesis: At Day 7 the proportion of decrease from baseline in the number of live lice in the Vamousse group does not exceed that in the Nix group. The distribution of the Day 0 to Day 7 change proportions deviated significantly from normality by the Shapiro-Wilk test for both the Vamousse and combined samples. However, the t-test is robust to such departures from normality for samples of this size and was used to compare the two groups on their mean change proportions; Test type: Superiority — The nonparametric Mann-Whitney test was also conducted to check on the effect of the non-normality of the change proportions. The null hypothesis is one-tailed. However, for consistency with the practice of reporting conservative p-values in clinical studies, the two-tailed p-value will be reported; p = .334, t-test, 2 sided — Alpha = .05 t: .976 df: 54 Mann-Whitney Z: 3.021 p(2-tailed) of Mann-Whitney Z: .003 Cohen's d = .294; Levine's test for violation of equality of variances nonsignificant; no df adjustment necessary; Mean Difference (Final Values) = .178, 95% CI 2-sided [-.187 to .543], Standard Error of Mean .182
Statistical Analysis 3: Comparison: Vamousse Spray 'n' Go vs Nix Creme Rinse Lice Treatment; Null hypothesis: At Day 14 the proportion of decrease from baseline in the number of live lice in the Vamousse group does not exceed that in the Nix group. The distribution of the Day 0 to Day 14 change proportion deviated significantly from normality by the Shapiro-Wilk test for both the Vamousse and combined samples. However, the t-test is robust to such departures from normality for samples of this size and was used to compare the two groups on the mean change proportions; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = .037, t-test, 2 sided — Alpha = .05 t: 2.276 df(adjusted, see comment below): 16.2 Mann-Whitney Z: 2.478 p(2-tailed) of Mann-Whitney Z: .013 Cohen's d = .947; Degrees of freedom for the t-test were adjusted for inequality of variances between the groups using the Satterthwaite correction: df(adj) = 16.2; Difference between proportions = .235, 95% CI 2-sided [.016 to .454], Standard Error of Mean .1034

ADVERSE EVENTS:
Time Frame: Day 0 through Day 14 for each participant.
Description: Systematic assessment was conducted by onsite clinical research staff members through collection of patient history, physical examination, and laboratory tests at baseline, Day 2, Day 7, and Day 14. This assessment was sufficiently thorough to have detected the onset or effects of any adverse reactions to the treatments and or excessive infestation due to insufficient mitigation by the treatments.
Arm/Group | Vamousse Spray 'n' Go | Nix Creme Rinse Lice Treatment
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/15
Other Adverse Events (participants affected / at risk) | 0/43 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/20/NCT05565820/Prot_SAP_000.pdf